CLINICAL TRIAL: NCT00327574
Title: Population Based Strategies for Effective Control of High Blood Pressure in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Wellcome Trust (Other); Imperial College London (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: GR 070854
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-05

CONDITIONS: Hypertension; Cardiovascular Disease; Obesity; Diabetes; Kidney Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Obesity; Diabetes Mellitus; Kidney Diseases

INTERVENTIONS:
Behavioral: Home heath education +/_ GP training

SUMMARY:
Studies have established that high blood pressure (BP) is the most common risk factor for cardiovascular disease (CVD). Despite a heavy burden of hypertension (33% of all persons aged 45 years and over), there are no reliable data on comparative strategies to manage hypertension in Pakistan. Our Wellcome Trust funded pilot study in Karachi, Pakistan on 320 adults aged 40 years and over showed that the prevalence of hypertension (95% CI) was 40.3% (34.9-45.7%), and CVD was 32.5% (27.6-37.8%).

We will now conduct a study with two components: 1) cross sectional study to determine the prevalence of CVD, and its determinants in Karachi, Pakistan; and 2) prospective, 2x2 factorial design, cluster allocation intervention study to evaluate the impact of a i) Population approach of household health education (HHE) by community health workers (CHW) on BP levels of population aged 5 years or over in low-middle income communities of Karachi; and ii) High-Risk approach of special BP management administered by intensively trained local general practitioners on BP levels of hypertensive subjects aged > = 40 years from the above population.

The cost effective BP control strategy would serve as a model for a much-needed national level hypertension control programme in Pakistan, and possibly other developing countries in South Asia.

We hypothesize that 1) HHE delivered by trained CHW is superior to no HHE in lowering BP levels of the population; and 2) management of hypertension by specially trained GPs is better than usual care provided in the communities of Karachi in lowering blood pressure of hypertensive subjects.

DETAILED DESCRIPTION:
The proposed study will be conducted among the low and middle-income population in Karachi. This population is likely to be particularly prone to CVD, has the poorest access to quality care, and is often prescribed expensive drugs by GPs.

Screening visit: The Community Health Workers (CHW) will pay home visits to invite all subjects aged 5 years or over to participate in the survey. The screening would have three levels: 1) Household screening for subjects aged 5 years and over (n= 17,850 individuals, 3000 households). 2) Adult screening for individuals aged 40 years or over (n= 4200 individuals). 3) Hypertensive adults screening (n= 1860 individuals) for those identified to have hypertension on adult screening will be invited for re-measurement of BP to confirm hypertension.

Intervention Effectiveness Study: This is a 2x2 factorial design, cluster allocation intervention study comparing controls with intervention by primary care GP, with or without health education. The main comparisons relate to the reduction of BP in a) all household members (aged > 5 years), and b) hypertensive adults (aged > 40 years).

Interventions: The sample will be assigned to four intervention groups:

* Group A: Routine care.
* Group B: Routine care plus Health Education
* Group C: Care provided by trained GP
* Group D: Care provided by trained GP plus Health Education.

ELIGIBILITY:
Inclusion Criteria:

* All subjects aged 5 years or over residing in randomly selected communities

Exclusion Criteria:

* Those who have severe co-morbid conditions
* Pregnancy
* Unable to give informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-06; Study Completion 2007-09

PRIMARY OUTCOMES:
Cross sectional: The prevalence (95% confidence intervals) of CVD, hypertension, diabetes, albuminuria, and mean values of lipid.
Intervention study: Changes in systolic and diastolic BP,
b) body mass index (BMI), e) waist hip ratio, and f) tobacco use from baseline to 2 year follow up visit
Cost Outcome Measures: These will be computed for hypertensive adults.
Primary outcomes: incremental cost per mm reduction in SBP, and DBP for each of the three intervention arms.
the three intervention arms

SECONDARY OUTCOMES:
Secondary Effect Outcomes: a) Proportion of subjects with mean follow-up BP less than 140/90 mm Hg,
and changes in b) BMI, c) waist hip ratio, and f) tobacco use.
Cost outcomes: the total cost per intervention and cost per subjects

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD MPH, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Jafar TH, Jafary FH, Jessani S, Chaturvedi N. Heart disease epidemic in Pakistan: women and men at equal risk. Am Heart J. 2005 Aug;150(2):221-6. doi: 10.1016/j.ahj.2004.09.025. PMID 16086922
- [Background] Jafar TH, Levey AS, Jafary FH, White F, Gul A, Rahbar MH, Khan AQ, Hattersley A, Schmid CH, Chaturvedi N. Ethnic subgroup differences in hypertension in Pakistan. J Hypertens. 2003 May;21(5):905-12. doi: 10.1097/00004872-200305000-00014. PMID 12714864
- [Derived] Jafar TH, Jehan I, Liang F, Barbier S, Islam M, Bux R, Khan AH, Nadkarni N, Poulter N, Chaturvedi N, Ebrahim S. Control of Blood Pressure and Risk Attenuation: Post Trial Follow-Up of Randomized Groups. PLoS One. 2015 Nov 5;10(11):e0140550. doi: 10.1371/journal.pone.0140550. eCollection 2015. PMID 26540210
- [Derived] Almas A, Jafar TH. Adiposity and blood pressure in South Asian children and adolescents in Karachi. Am J Hypertens. 2011 Aug;24(8):876-80. doi: 10.1038/ajh.2011.67. Epub 2011 Apr 21. PMID 21509050
- [Derived] Jafar TH, Islam M, Hatcher J, Hashmi S, Bux R, Khan A, Poulter N, Badruddin S, Chaturvedi N; Hypertension Research Group. Community based lifestyle intervention for blood pressure reduction in children and young adults in developing country: cluster randomised controlled trial. BMJ. 2010 Jun 7;340:c2641. doi: 10.1136/bmj.c2641. PMID 20530082
- [Derived] Jafar TH, Hatcher J, Poulter N, Islam M, Hashmi S, Qadri Z, Bux R, Khan A, Jafary FH, Hameed A, Khan A, Badruddin SH, Chaturvedi N; Hypertension Research Group. Community-based interventions to promote blood pressure control in a developing country: a cluster randomized trial. Ann Intern Med. 2009 Nov 3;151(9):593-601. doi: 10.7326/0003-4819-151-9-200911030-00004. PMID 19884620
- [Derived] Jafar TH, Qadri Z, Chaturvedi N. Coronary artery disease epidemic in Pakistan: more electrocardiographic evidence of ischaemia in women than in men. Heart. 2008 Apr;94(4):408-13. doi: 10.1136/hrt.2007.120774. Epub 2007 Jul 23. PMID 17646192